CLINICAL TRIAL: NCT06784219
Title: Development and Validation of Self-Reported Surveillance Questionnaire of Periodontal Health in Indian Population
Status: Not yet recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Other Study IDs: ADITIPERIO(SURVEILLENCE)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients seeking dental care: A cross-sectional study based on a convenience sample of consecutive patients seeking dental care at the Post Graduate Institute of Dental Sciences, Rohtak. The participants will comprise of individuals aged 18 or above. The exclusion criteria are: 1) edentulous adults, 2) pregnant females, 3) individuals having received antibiotic medication within the previous 3 months, 4) individuals having received professional periodontal treatment within the previous 12 months.
  Interventions: Diagnostic Test: Hindi version of self reported oral health questionnaire

INTERVENTIONS:
Diagnostic Test: Hindi version of self reported oral health questionnaire — The original 8-item CDC/AAP questionnaire as well as other selected periodontal disease surveillance questions will be translated into Hindi through forward translation, backward translation, and expert committee process to reach a consensus and produce a prefinal version. The prefinal version questionnaire will be pilot tested on a sample of 20 patients to evaluate the overall comprehension by non-professionals. On the basis of responses and evaluation from the participants, the questionnaire will be further refined to build the final version. The final version of the questionnaire will be administered to patients seeking care from out-patient department of department of Periodontics at PGIDS, Rohtak. The participants will be required to fill the questionnaire by themselves prior to periodontal examination, without any help from others.

SUMMARY:
Rationale- Periodontal disease is a dynamic inflammatory condition, that affects the periodontium and has a profound effect on the overall systemic health of the individual. Unfortunately, the symptoms of periodontal disease often go unnoticed by affected individuals and this contributes towards unpleasant and irreversible consequences such as tooth loss. Hence it is important to develop an easy, cost effective and widely acceptable method for the patients to assess their periodontal health.

Objectives- To translate, culturally adapt and validate the CDC/AAP questionnaire along with other relevant surveillance questions in the Hindi language according to the new case definitions of periodontal diseases.

Methods- The original 8-item CDC/AAP questionnaire as well as other selected periodontal disease surveillance questions will be translated into Hindi through forward translation, backward translation, and expert committee process to reach a consensus and produce a final version. The final version of the questionnaire will be administered to patients seeking care from out-patient department of department of Periodontics at PGIDS, Rohtak. Full-mouth periodontal examination, consisting of measurements of the probing pocket depth (PPD), full mouth bleeding score (FMBS) and clinical attachment level (CAL) at six sites per tooth using periodontal probe will be carried out for each participant.

DETAILED DESCRIPTION:
Background- Periodontal disease, with its chronic systemic effects and poor influence on the quality of life of the patient, is global healthcare challenge. Hence there is a for timely diagnosis and treatment of the patients.

Rationale- Periodontal disease is a dynamic inflammatory condition, that affects the periodontium and has a profound effect on the overall systemic health of the individual. Unfortunately, the symptoms of periodontal disease often go unnoticed by affected individuals and this contributes towards unpleasant and irreversible consequences such as tooth loss. Hence it is important to develop an easy, cost effective and widely acceptable method for the patients to assess their periodontal health.

Objectives- To translate, culturally adapt and validate the CDC/AAP questionnaire along with other relevant surveillance questions in the Hindi language according to the new case definitions of periodontal diseases.

Methods- The original 8-item CDC/AAP questionnaire as well as other selected periodontal disease surveillance questions will be translated into Hindi through forward translation, backward translation, and expert committee process to reach a consensus and produce a final version. The final version of the questionnaire will be administered to patients seeking care from out-patient department of department of Periodontics at PGIDS, Rohtak. Full-mouth periodontal examination, consisting of measurements of the probing pocket depth (PPD), full mouth bleeding score (FMBS) and clinical attachment level (CAL) at six sites per tooth using periodontal probe will be carried out for each participant.

Expected outcomes- Response to self- reported questionnaire (individual questions as well as in combination) in Hindi speaking population and its ability to predict periodontal status will be evaluated. If found to be valid, this could serve as a vital tool for periodontal health screening for Hindi speaking population at the primary care level.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or above and voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Edentulous adults Pregnant females Individuals having received antibiotic medication within the previous 3 months Individuals having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study has been designed as a cross-sectional study based on a convenience sample of consecutive patients seeking dental care at the Post Graduate Institute of Dental Sciences (PGIDS), Rohtak. The participants will comprise of individuals aged 18 or above and voluntarily agreeing to participate in the study. The exclusion criteria are: 1) edentulous adults, 2) pregnant females, 3) individuals having received antibiotic medication within the previous 3 months, 4) individuals having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months. Informed consent will be obtained from each participant prior to enrolment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Response to self- reported questionnaire (individual questions as well as in combination) in Hindi speaking population. | 1-1.5 months
  Hindi version of self-reported oral health questionnaire will be administered to consecutive patients attending out-patient department. Periodontal status of the patients was then evaluated by measuring PI, GI, PPD, BOP, CAL. Their responses were then correlated with the periodontal status.

SECONDARY OUTCOMES:
Correlation of responses of Self-Reported Questionnaire for periodontal health with demographic data of the patient | 1-1.5 months
  The responses will be evaluated along with demographic data of the patient like age, gender, level of education, occupation, marital status and place of residence
Correlation of Bleeding on probing (BOP) with response of Self- Reported Questionnaire for periodontal health | 1-1.5 months
  Bleeding on probing was checked for each patient and response from their Hindi version self-reported oral health questionnaire were correlated
Correlation of Probing pocket depth (PPD) with Self-Reported Questionnaire for periodontal health | 1-1.5 months
  Probing pocket depth was measured for each patient and their response of the Hindi version self-reported questionnaire was correlated
Correlation of Clinical attachment level (CAL) with Self-Reported Questionnaire for periodontal health | 1-1.5 months
  Clinical attachment loss was measured for each patient and their response of the Hindi version of self-reported oral health questionnaire was correlated

CONTACTS AND LOCATIONS:
Overall Officials: Aditi SANGWAN, Principal Investigator — Post graduate institute of Dental Sciences ROHTAK; RINDA SHARMA, Principal Investigator — PT. B. D. SHARMA UHSR HARYANA
Locations (1):
- Post Graduate Institute O Fdental Sciences, Rohtak, Haryana, India